CLINICAL TRIAL: NCT01983930
Title: Memory Training Versus Yogic Meditation Training in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-000821
Record Dates: First submitted 2013-10-30; First posted 2013-11-14 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2017-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory impairment; Meditation; Yoga; memory training; Mild cognitive impairment; MCI; geriatric; fMRI
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders | interventions — Meditation; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memory Training (Active Comparator): Group memory training will be administered for amnestic mild cognitive impairment (MCI)
  Interventions: Behavioral: Memory Training
- Kundalini yoga and meditation (Experimental): Participants will engage in weekly yoga classes and daily 20 minute meditation
  Interventions: Behavioral: Kundalini yoga and meditation

INTERVENTIONS:
Behavioral: Kundalini yoga and meditation — Participants will participate in a 60 minute yoga and meditation session weekly for 12 weeks and will be assigned a daily Kirtan Kriya meditation (12 minute duration) for 12 weeks.
  Arms: Kundalini yoga and meditation
Behavioral: Memory Training — Participants will attend a weekly memory training class for 12 weeks as well as receive daily memory homework (12 minute duration) for the 12 weeks.
  Arms: Memory Training

SUMMARY:
The purpose of this pilot study is to test whether 6 months of supervised weekly Kundalini yoga classes and a brief daily meditation homework assignment can improve memory and thinking in older adults with mild memory complaints when compared to weekly classes of memory training with daily homework assignments.

DETAILED DESCRIPTION:
The purpose of this pilot study intervention is to investigate brain mechanisms of response to memory enhancement training (MET) compared to Kundalini yoga and "Kirtan Kriya" meditation using functional magnetic resonance imaging (fMRI) that will be acquired from each subject at baseline and at 12 weeks (post-randomization).

Overall, the investigators anticipate recruiting 66 adults with memory complaints and diagnosed with MCI for adults 55 years old and older. Subjects will either receive: (1) MET class for 60 minutes per week; or (2) Kundalini yoga and "Kirtan Kriya" meditation class for 60 minutes per week. All assessments will be completed immediately after the interventions for a total of 10 visits in 12 weeks and a follow-up visit at 6 months (24 weeks)to monitor the overall benefit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment amnestic type
* Clinical Dementia Rating scale score of 0.5
* SufficientEnglish proficiency and 8th grade or higher reading level as determined by the word reading subtest of the Wide Range Achievement Test-IV
* Capacity to provide informed consent.

Exclusion criteria:

* Any current or past psychiatric disorders, or recent unstable medical or neurological disorders
* Any disabilities preventing their participation in the memory enhancement training (MET) (e.g. severe visual or hearing impairment)
* Insufficient English proficiency
* Diagnosis of dementia
* Mini Mental Health Examination score of 24 and below
* Psychoactive medications
* Participation in a psychotherapy that involves cognitive training
* Do not meet criteria for Mild cognitive impairment subtype
* Prior or current training in yoga.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, MD, MS, Principal Investigator — UCLA Semel Institute
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eyre HA, Siddarth P, Acevedo B, Van Dyk K, Paholpak P, Ercoli L, St Cyr N, Yang H, Khalsa DS, Lavretsky H. A randomized controlled trial of Kundalini yoga in mild cognitive impairment. Int Psychogeriatr. 2017 Apr;29(4):557-567. doi: 10.1017/S1041610216002155. Epub 2017 Jan 16. PMID 28088925

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single site outpatient clinic in the U.S.
Pre-assignment Details: 168 volunteers were assessed for eligibility, of which 51 declined to participate and 32 did not meet inclusion criteria. Eighty-five volunteers consented to participate, of which 81 passed screening and were enrolled; two of 81 enrolled participants withdrew post-randomization and did not receive the allocated intervention.
Groups:
- Memory Training: Group memory training will be administered for amnestic MCI
  Memory Training: Participants will attend a weekly memory training class for 12 weeks as well as receive daily memory homework (12 minute duration) for the 12 weeks.
Period: Overall Study
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Started | 41 | 38
Completed | 32 | 29
Not Completed | 9 | 9
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memory Training | Kundalini Yoga and Meditation | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.7) | 67.6 (8.0) | 67.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 30 | 24 | 54
  Non-Caucasian | 11 | 14 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Measures - Hopkins Verbal Learning Test (HVLT) Total Recall Score
Description: Primary outcome measures were administered by a cognitive battery of neuropsychological and included memory and executive functioning. Verbal memory was measured with the Hopkins Verbal Learning Test (HVLT) total recall scores. The HVLT form contains 12 nouns, four words each from one of three semantic categories (e.g., precious gems, articles of clothing, vegetables, etc.), to be learned over the course of three learning trials. When scoring the HVLT, the three learning trials are combined to calculate a total recall score. Total scores range from 0-36 with higher scores indicating better outcome.
Time Frame: At baseline and at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memory Training: Group memory training will be administered for amnestic MCI.
  Memory Training: Participants will attend a weekly memory training class for 12 weeks as well as receive daily memory homework (12 minute duration) for the 12 weeks.
- Kundalini Yoga and Meditation: Participants will engage in weekly yoga classes and daily 20 minute meditation.
  Kundalini yoga and meditation: Participants will participate in a 60 minute yoga and meditation session weekly for 12 weeks and will be assigned a daily "Kirtan Kriya" meditation (12 minute duration) for 12 weeks.
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 41 | 38
units on a scale
  Baseline | 26.02 (5.42) | 25.76 (6.20)
  6 Months | 27.96 (5.44) | 28.81 (6.52)

2. Secondary Outcome: Clinical Global Impression Scale
Description: The CGI measures severity of illness and global improvement. The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI global improvement scores range from 1 (very much improved) through to 7 (very much worse).
Time Frame: Baseline, weeks 2, 4, 6, 8, 10, 12, 24
Population: Data were not collected.
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: Secondary outcomes measures included mood assessments with the GDS, a self-assessment scale often used in geriatric depression trials. The GDS is a 30-item screening tool used to identify depression in older adults. In scoring the Geriatric Depression Scale, each item is scored 0 or 1. The total score on the scale ranges from 0 to 30 with higher scores indicating worse outcome.
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 41 | 38
units on a scale
  Baseline | 5.7 (5.6) | 7.5 (5.1)
  Week 24 | 3.2 (2.5) | 3.9 (2.5)

4. Secondary Outcome: Change in Functional Magnetic Resonance Imaging (fMRI) Connectivity
Description: FMRI scans will be obtained at baseline and after 12 weeks follow up. Default mode network findings were analyzed and significant effects were identified for yoga and memory enhancement training groups.
Time Frame: 12 weeks
Measure: Number; unit: p-value
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Number analyzed (Participants) | 11 | 14
p-value
  pregenual anterior cingulate cortex (ACC) p-value | 0.011 | 0.001
  frontal medial cortex (FMC) p-value | 0.035 | 0.001

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Memory Training | Kundalini Yoga and Meditation
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No